CLINICAL TRIAL: NCT07259148
Title: Non-Inferiority Randomized Clinical Trial Comparing Behavioral Therapy Plus Pharmacotherapy Versus Pelvic Floor Muscle Training Plus Pharmacotherapy in Women With Urgency Urinary Incontinence
Brief Title: Behavioral Interventions Versus Pelvic Floor Muscle Therapy as Adjuncts to Anticholinergic Pharmacotherapy for Urgency Urinary Incontinence: A Non-Inferiority Trial
Acronym: NI-UUI-2025
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emilio José Dávila Álvarez (Other)
Collaborators: Hospital Militar Escuela "Dr. Alejandro Dávila Bolaños" (Other)
Responsible Party: Sponsor-Investigator, Emilio José Dávila Álvarez, Sponsor-Investigator / Principal Investigator, Hospital Militar Escuela "Dr. Alejandro Dávila Bolaños"
Organization: Hospital Militar Escuela "Dr. Alejandro Dávila Bolaños" (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HMEADB-IUU-2025
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Urgency Urinary Incontinence
Keywords: Urgency urinary incontinence; Overactive bladder; Pelvic floor muscle therapy; Behavioral therapy; Bladder training; Anticholinergic pharmacotherapy; Oxibutinine; Mirabegron; Non-inferiority trial; Women's health
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — oxybutynin; mirabegron

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel-group, randomized controlled trial comparing pelvic floor muscle therapy versus behavioral therapy, both as adjuncts to standardized anticholinergic pharmacotherapy.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors and statisticians will be blinded to group allocation. Participants and care providers cannot be blinded due to the nature of the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic Floor Muscle Therapy + Pharmacotherapy (Active Comparator): Supervised pelvic floor muscle training (PFMT) twice weekly for 8 weeks, including slow and fast contractions, posture education, and home exercises. Combined with standardized pharmacotherapy: oxybutynin 5 mg every 12 hours; switch to mirabegron 25-50 mg daily if adverse effects or insufficient response occur.
  Interventions: Behavioral: Pelvic Floor Muscle Training (PFMT); Drug: Oxybutynin / Mirabegron (Standardized Pharmacotherapy)
- Behavioral Therapy + Pharmacotherapy (Active Comparator): Behavioral intervention consisting of bladder training, fluid management, reduction of bladder irritants, sleep hygiene, and healthy lifestyle counseling. Combined with standardized pharmacotherapy: oxybutynin 5 mg every 12 hours; switch to mirabegron 25-50 mg daily if adverse effects or insufficient response occur.
  Interventions: Behavioral: Behavioral Bladder Training Program; Drug: Oxybutynin / Mirabegron (Standardized Pharmacotherapy)

INTERVENTIONS:
Behavioral: Pelvic Floor Muscle Training (PFMT) — Supervised pelvic floor muscle training twice weekly for 8 weeks, including 3 sets of slow contractions (6-8 seconds) and 3 sets of fast contractions, posture education, breathing training, and daily home exercises.
  Arms: Pelvic Floor Muscle Therapy + Pharmacotherapy
Behavioral: Behavioral Bladder Training Program — Structured behavioral program including timed voiding every 2 hours with weekly interval increases, suppression of urgency techniques, fluid optimization, reduction of bladder irritants, sleep hygiene measures, and lifestyle recommendations.
  Arms: Behavioral Therapy + Pharmacotherapy
Drug: Oxybutynin / Mirabegron (Standardized Pharmacotherapy) — Oxybutynin 5 mg every 12 hours as first-line therapy. Mirabegron 25-50 mg daily will be used in cases of intolerance or inadequate response. Medication use will be monitored and recorded.

SUMMARY:
Urgency urinary incontinence (UUI) is a common condition that significantly affects women's quality of life. Pharmacotherapy is often used as first-line treatment, but its effectiveness can be limited unless combined with non-pharmacological interventions. Pelvic floor muscle therapy (PFMT) is widely recommended; however, access to specialized physiotherapy services is limited in many low-resource settings such as Nicaragua. Behavioral interventions-including bladder training, fluid control, avoidance of bladder irritants, and sleep-hygiene strategies-represent a low-cost alternative, but direct comparative evidence against PFMT is limited.

This randomized, controlled, non-inferiority clinical trial will compare two adjuvant strategies combined with standard anticholinergic pharmacotherapy (oxibutinine):

1. Pelvic floor muscle therapy (PFMT), and
2. Behavioral interventions (bladder training and lifestyle modification).

Eighty adult women with urgency urinary incontinence or mixed incontinence with urgency-predominance will be randomized 1:1. The intervention period is 8 weeks, with assessments at baseline, week 4, week 8, and an exploratory follow-up at week 12.

The primary outcome is the change in the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) score from baseline to week 8. A non-inferiority margin of 3 points will be applied. Secondary outcomes include episodes of urgency/incontinence per 24 h, ICIQ-LUTSqol scores, patient-reported global improvement (PGI-I), adherence, and adverse events.

This study aims to determine whether behavioral interventions are not inferior to PFMT as adjuncts to pharmacotherapy, potentially offering a feasible and more accessible therapeutic alternative for women with UUI in resource-limited healthcare environments.

DETAILED DESCRIPTION:
Urgency urinary incontinence (UUI) is highly prevalent among women and is associated with substantial psychosocial, functional, and economic consequences. Although anticholinergic medications are commonly used, their effectiveness is often improved when combined with adjunctive non-pharmacological interventions. Pelvic floor muscle therapy (PFMT) has strong evidence supporting its use; however, its implementation requires trained personnel, scheduled sessions, and specialized infrastructure, which may not be accessible in low-resource settings.

Behavioral interventions-including bladder training, fluid management, avoidance of bladder irritants, dietary modifications, bowel regulation, and sleep-hygiene measures-represent a practical and low-cost alternative. Despite their clinical utility, there is limited evidence from randomized trials directly comparing behavioral interventions to PFMT when used as adjuncts to pharmacotherapy.

This study is a randomized, controlled, non-inferiority trial conducted at a national reference hospital in Nicaragua. The trial will enroll 80 adult women (≥18 years) diagnosed with UUI or mixed urinary incontinence with urgency predominance. Participants will be randomized in a 1:1 ratio to receive either (1) PFMT plus pharmacotherapy or (2) behavioral interventions plus pharmacotherapy. Oxibutinine (5 mg every 12 hours) will be used as the standard pharmacological agent, with mirabegron available as second-line therapy when intolerance occurs.

The intervention period lasts 8 weeks. PFMT includes supervised sessions twice per week plus a structured home-exercise program. Behavioral interventions include individualized bladder-training schedules, fluid-intake monitoring, avoidance of irritants, lifestyle counseling, and sleep-hygiene strategies. Adherence will be monitored at weeks 4 and 8.

The primary outcome is the change in ICIQ-SF score from baseline to week 8, with non-inferiority defined as an upper bound of the 95% confidence interval below 3 points. Secondary outcomes include ICIQ-LUTSqol, episodes of urgency and incontinence (3-day bladder diary), PGI-I, adherence to interventions, and adverse events. Week 12 assessments will explore persistence of clinical benefit.

This study is designed to generate locally applicable evidence to inform clinical practice in settings where PFMT availability is limited. Demonstrating non-inferiority of behavioral interventions could support more accessible and cost-effective management strategies for women with UUI.

ELIGIBILITY:
Inclusion Criteria

* Women aged ≥18 years.
* Symptoms of urgency urinary incontinence (UUI) or mixed urinary incontinence with predominance of urgency, with duration ≥3 months.
* Clinical diagnosis of UUI based on history, physical examination, and a 3-day bladder diary.
* Predominance of urgency defined as: at least 50% of total recorded episodes in the bladder diary correspond to urgency (with or without leakage).
* Baseline ICIQ-SF score ≥6.
* Ability to attend scheduled visits and comply with assigned intervention.
* Signed informed consent.

Exclusion Criteria:

* Pure stress urinary incontinence.
* Mixed urinary incontinence with predominance of stress defined as: more than 70% of episodes in the 3-day bladder diary are triggered by physical effort.
* Symptomatic advanced pelvic organ prolapse (POP-Q stage ≥III).
* Active or recent urinary tract infection (within the last 7 days).
* Prior use of anticholinergics or β3-agonists that cannot be discontinued for a 14-day washout period.
* Pregnancy or breastfeeding.
* Neurological or psychiatric disorders affecting bladder function, record-keeping, or adherence.
* Cognitive or functional difficulty preventing understanding or completion of study procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female participants only, due to the epidemiology and pathophysiology of urgency urinary incontinence in women.
Enrollment: 80 (Estimated)
Dates: Start 2025-11-22 (Actual); Primary Completion 2026-01-23 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in ICIQ-SF Total Score from Baseline to Week 8 | Baseline and Week 8
  This measure evaluates the change in the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) total score between baseline and week 8. The ICIQ-SF assesses frequency, severity, and impact of urinary incontinence on quality of life. Scores range from 0 to 21, with higher scores indicating greater severity.

SECONDARY OUTCOMES:
Change in ICIQ-LUTSqol Score from Baseline to Week 8 | Baseline and Week 8
  This measure evaluates the change in the International Consultation on Incontinence Questionnaire-Lower Urinary Tract Symptoms Quality of Life (ICIQ-LUTSqol) score between baseline and week 8. The questionnaire assesses the impact of urinary incontinence on daily activities, psychological well-being, and social functioning. Total scores range from 19 to 76, with higher scores indicating greater impairment.
Change in Number of Urgency Urinary Incontinence Episodes per 24 Hours | Baseline and Week 8
  Change in the frequency of urgency urinary incontinence episodes per 24 hours, based on a 3-day bladder diary completed at baseline and week 8.
Patient Global Impression of Improvement (PGI-I) at Week 8 | Week 8
  The PGI-I is a validated single-item global rating scale in which participants rate their improvement on a 7-point scale ranging from "very much better" to "very much worse." Lower scores indicate greater subjective improvement.
Change in Number of Micturitions per 24 Hours | Baseline and Week 8
  Change in the total number of micturitions per 24 hours, based on a 3-day bladder diary completed at baseline and week 8.
Change in Number of Urgency Urinary Incontinence Episodes per 24 Hours | Baseline and Week 8
  Change in the frequency of urgency urinary incontinence episodes per 24 hours, recorded in a 3-day bladder diary at baseline and week 8.
Change in Number of Urgency Episodes per 24 Hours | Baseline and Week 8
  Change in the number of urgency episodes per 24 hours, obtained from a 3-day bladder diary at baseline and week 8.
Change in Number of Absorbent Pads Used per 24 Hours | Baseline and Week 8
  Change in the total number of absorbent pads used per 24 hours, as documented in a 3-day bladder diary at baseline and week 8.
Adherence to Assigned Intervention | Throughout the 8-week intervention period
  Proportion of participants achieving ≥80% adherence to the assigned intervention protocol, monitored through weekly checklists and session attendance logs.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Militar Escuela Dr. Alejandro Dávila Bolaños, Managua, Managua Department, Nicaragua

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect participant privacy and based on institutional policy. Summary aggregated results will be reported in ClinicalTrials.gov according to regulatory requirements.